CLINICAL TRIAL: NCT04324762
Title: De-Implementation Of Routine Chest Radiographs After Adoption of Ultrasound Guided Insertion and Confirmation of Central Venous Catheter Protocol
Brief Title: Implementation of Ultrasound Guided Central Venous Catheter Confirmation Protocol
Acronym: DRAUP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201807001
Record Dates: First submitted 2020-03-20; First posted 2020-03-27 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Behavior; Process, Acceptance; Inertia of Accommodation
Keywords: ultrasound; central venous catheter; POCUS; chest radiography; Dissemination & Implementation; De-Implementation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: targetted implementation strategies — strategies at the individual and institutional level to promote implementation of an evidenced based innovation and de-implementation of an unnecessary, low value diagnostic test.

SUMMARY:
The bedside use of ultrasound after central venous catheter (CVCs) insertion has lagged behind other applications in medicine, thus presenting an opportunity for innovative, evidence-based research that will influence clinician behavior. This research focuses on bedside ultrasound applications as an example, to evaluate clinical practice change. Chest radiographs are associated with delays in initiating time-critical interventions and present an unexamined opportunity for improving patient care by evaluating the use of ultrasound in lieu of chest radiographs after CVC insertion. Strategic interventions for implementation are needed to hasten the adoption of this clinical innovation (ultrasound guided CVC confirmation protocol) allowing them to de-implement chest xrays when no longer indicated.

DETAILED DESCRIPTION:
The placement of central venous catheters (CVCs) is a common procedure performed in critically ill patients, with millions placed annually. The routine use of chest radiographs for CVC confirmation is outdated. Chest radiographs are associated with delays in initiating time-critical interventions and present an unexamined opportunity for improving resource utilization and associated costs. Radiography has been used for over 50 years for this purpose in the absence of other options. Emerging evidence suggests that a post-procedure chest radiographs are unnecessary when ultrasound is used to confirm catheter position and exclude pneumothorax (PCEP). Yet few in the medical community are likely aware of these data and even among those who are aware, chest radiographs continues to be the routine modality used for CVC PCEP.

The average 17 years it takes to translate clinical research into practice is too long and presents an opportunity to expedite implementation of innovations in critical care medicine. For the proposed project, "De-Implementation Of Routine Chest Radiographs After Adoption of Ultrasound Guided Insertion and Confirmation of Central Venous Catheter Protocol (DRAUP)", the hypothesis is that identifying determinants of behavior for intervention development (Aim 1) will increase the likelihood of developing successful strategies that will yield faster clinical adoption. Understanding the behavioral adaptations that have to occur is key to developing strategies that increase the uptake of evidence into healthcare practice and improving health outcomes. These strategies (targeting adoption and substitution) will then be implemented in a local Emergency Department (Aim 2) to determine if these selected implementation strategies will increase provider adoption, fidelity, and organizational penetrance (Aim 3) of ultrasound-guided CVC PCEP. A good clinical outcome would be a decrease in provider dependence on chest radiographs after ultrasound-guided CVC PCEP.

ELIGIBILITY:
Inclusion Criteria:

* have a clinical role in the placement and maintenance of central venous catheters

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical healthcare workers involved in the placement and/or maintenance of central venous catheters (nurses, doctors, administrators)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adoption | 1 year
  Adoption will be measured by calculating the absolute number and proportion who utilize POCUS guided protocol and deimplement chest radiographs after central venous catheter placement
De-adoption | 1 year
  De-adoption will be measured by calculating the absolute number and proportion who do not obtain chest radiographs after central venous catheter placement
Fidelity | 1 year
  Fidelity will be measured by calculating the degree (%) to which the DRAUP algorithm was implemented as it was prescribed

SECONDARY OUTCOMES:
Effectiveness | 1 year
  Effectiveness will be measured by calculating the sensitivity/specificity of POCUS guided CVC confirmation

CONTACTS AND LOCATIONS:
Overall Officials: Enyo A Ablordeppey, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington Unversity School Of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared via manuscript publication; specific IPDs can be requested by email. All shared data will be in the form of group assessments as to not identify an individual response or behavior pattern.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months (timeline for anticipated study protocol manuscript)

REFERENCES:
- [Derived] Ablordeppey EA, Powell B, McKay V, Keating S, James A, Carpenter C, Kollef M, Griffey R. Protocol for DRAUP: a deimplementation programme to decrease routine chest radiographs after central venous catheter insertion. BMJ Open Qual. 2021 Oct;10(4):e001222. doi: 10.1136/bmjoq-2020-001222. PMID 34663588